CLINICAL TRIAL: NCT00540917
Title: Phase II Clinical Trial is to Compare Epidermal Temperature Measurements During 1.Laser Treatment at Standard Treatment Energies 2.Cryogen Spray Cooling (CSC) Plus Laser Treatment. 3.Contact Cooling Plus Laser Treatment.
Brief Title: Measurement Skin Temperature During Pulsed Laser Exposure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other); Candela Corporation (Industry)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, J S Nelson, M.D., Ph.D.,Professor of Surgery and Biomedical Engineering, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19992250
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cooling spray (Experimental): cooling spray during laser treatment
  Interventions: Procedure: cooling spray during laser treatment

INTERVENTIONS:
Procedure: cooling spray during laser treatment — skin temperature measurement
  Other Names: laser treatment

SUMMARY:
Lasers are the treatment modality of choice for Port Wine Stain birthmarks.The epidermis is not totally spared due to partial absorption of energy therein by melanin that presents an optical barrier through which the light must pass to reach the underlying blood vessels. Absorption of laser energy by melanin causes localized heating in the epidermis, which may, if not controlled, produce permanent complications such as hypertrophic scarring or dyspigmentation.

DETAILED DESCRIPTION:
The researchers want to establish a correlation between non-invasive skin temperature measurements and the minimum laser energy during skin laser treatment using cryogen spray cooling.

This study would eliminate the need for test pulses to estimate the safe and acceptable radiant exposure prior to laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* 7 years of age and older with diagnosis of port wine stain birthmark
* 18 years of age and older with no port wine stain
* non-pregnant women
* apparent good health

Exclusion Criteria:

* age less than 7 years old
* pregnant women
* history of photodermatoses or skin cancer
* current use of photosensitizing drugs

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2002-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
skin temperature during laser treatment | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: John S. Nelson, M.D., Ph.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical Clinic University of California Irvine, Irvine, California, United States